CLINICAL TRIAL: NCT05150275
Title: Retrospective Study Comparing Classic Vaginal Hysterectomy to vNOTES Hysterectomy
Brief Title: Study Comparing Classic Vaginal Hysterectomy to vNOTES Hysterectomy
Acronym: H-vNOTES
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8418
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Hysterotomy
Keywords: Hysterotomy; vNOTES; Laparoscopy; Vaginal route

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
vNOTES is a new surgical approach that has been used for less than 10 years. Several studies compare it to laparoscopy but none compare it to the classic vaginal route.

The aim of the research is to analyze postoperative pain

ELIGIBILITY:
Inclusion criteria:

* Adult woman (≥18 years old)
* Woman having undergone a vaginal hysterectomy and by vNOTES at Strasbourg University Hospitals between 01/01/2017 and 05/31/2021
* Woman who did not express her opposition to the reuse of her data for the purposes of this research.

Exclusion criteria:

* Woman who expressed her opposition to participating in the study
* Surgical procedure associated with hysterectomy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult woman having undergone a vaginal hysterectomy and by vNOTES at Strasbourg University Hospitals between 01/01/2017 and 05/31/2021
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Analysis of postoperative pain in patients who have had a vaginal hysterectomy | Files analysed retrospectively from January 01, 2017 to May 31, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GARBIN, MD, Principal Investigator — Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de chirurgie gynécologique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France